CLINICAL TRIAL: NCT01881958
Title: The Safety and Efficacy of Administrating DiaPep277® Vaccination in Type 1 Diabetes Patients.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the manufacturer decided to halt manufacturing the vaccine
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0224-13-HMO-CTIL
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Type One Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DiaPep277® (Experimental)
  Interventions: Drug: DiaPep277®

INTERVENTIONS:
Drug: DiaPep277®

SUMMARY:
Type 1 diabetes is caused by an autoimmune process resulting in a selective destruction of the pancreatic insulin-secreting beta-cell. DiaPep277® is a small, lyophilized powder containing 24 Amino-acids. We have proved in former studies that DiaPep277® can slow down beta cells destruction in the pancreas and therefore decelerate the progress of Diabetes.

The objective of the study is to assess the efficacy and safety of administrating DiaPep277® in type 1 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting C-peptide levels >= 0.2nmol/L.
2. Diagnosis of type 1 diabetes
3. No pregnancies or planned pregnancies of female subjects

Exclusion Criteria:

1. The subject has any significant diseases or conditions, including psychiatric disorders and substance abuse that, in the opinion of the Investigator, are likely to affect the subject's response to treatment or the ability to complete the study.
2. The subject has a history of any kind of malignant tumor (not including basal cell skin cancer).
3. The subject has clinical evidence of any diabetes-related complication that in the opinion of the Investigator would interfere with the subject's participation in and/or completion of the study.
4. Subject has history of endogenous allergic reactivity:

   * Severe allergic reaction or severe exacerbation of allergic asthma within 12 months prior to the Screening-Ext Visit.
   * Ongoing systemic asthma treatment.
   * Subjects with history of life threatening or severe allergy, re-occurrence of which cannot be ruled out based on the Investigator's judgment.
5. The subject has known allergy to lipid emulsions.
6. The subject has a known immune deficiency from any disease, or a condition associated with an immune deficiency.
7. The subject is receiving immunosuppressive or immunomodulating agents or cytotoxic therapy or any medication that in the opinion of the Investigator might interfere with the study.
8. The subject has any of the following clinically significant laboratory abnormalities:

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of the normal (ULN) at the Screening-Ext Visit.
   * Total bilirubin greater than 1.3 times the ULN at the Screening-Ext Visit.
   * Subjects with severe renal failure at the Screening-Ext visit (as defined by glomerular filtration rate < 30 mL/min/1.73 m2 by Cockroft und Gault calculation • Clinically significant laboratory abnormalities, confirmed by repeat measurement, which may interfere with the assessment of safety and / or efficacy of the study drug, other than hyperglycemia and glycosuria at the Screening-Ext Visit.
   * Fasting triglycerides <1000 mg/dL (11.3 mmol/L) at the Screening-Ext Visit. Suitable medical therapy for treatment of hyperlipidemia is allowed.
9. The subject is a known or suspected drug abuser.
10. The subject is known to test positive for HIV antibodies.
11. The subject has chronic hematologic disease.
12. The subject has liver disease such as cirrhosis or chronic active hepatitis.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Estimated); Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
efficacy will be measured by comparing Hemoglobin A1c | two years

SECONDARY OUTCOMES:
Safety will be evaluated calculating number of Adverse Events. | two years